CLINICAL TRIAL: NCT04633135
Title: Research on Emissions, Air Quality, Climate and Cooking Technologies in Northern Ghana
Acronym: REACCTING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Boulder (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency); U.S. National Science Foundation (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Hannigan, Principle Investigator, University of Colorado, Boulder
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: REACCTING; GEO-1211668 (Other Grant/Funding Number: NSF); RD-8354201 (Other Grant/Funding Number: EPA)
Record Dates: First submitted 2020-09-14; First posted 2020-11-18 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Inflammation; Growth Retardation
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Intervention Model Description: There were 4 groups, 3 intervention and 1 control, all operating over the same period.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control (No Intervention): Households enrolled in the control arm of the study did not receive either improved cookstove
- Gyapa/Gyapa (Experimental): Households enrolled in the Gyapa/Gyapa arm of the study received two Gyapa stoves for free
  Interventions: Device: Gyapa stove
- Gyapa/Philips (Experimental): Households enrolled in the Gyapa/Philips arm of the study received one Gyapa stove and one Philips stove for free
  Interventions: Device: Philips stove; Device: Gyapa stove
- Philips/Philips (Experimental): Households enrolled in the Philips/Philips arm of the study received two Philips stoves for free
  Interventions: Device: Philips stove

INTERVENTIONS:
Device: Philips stove — Philips Smokeless stove HD4012LS
  Other Names: Gasifier stove
  Arms: Gyapa/Philips; Philips/Philips
Device: Gyapa stove — Wood stove made in Ghana
  Other Names: Rocket stove
  Arms: Gyapa/Gyapa; Gyapa/Philips

SUMMARY:
REACCTING (Research on Emissions, Air quality, Climate, and Cooking Technologies in Northern Ghana) is an interdisciplinary randomized cookstove intervention study in the Kassena-Nankana District of Northern Ghana. The study tests two types of biomass burning stoves that have the potential to meet local cooking needs and represent different "rungs" in the cookstove technology ladder: a locally-made, low-tech Gyapa rocket stove and the imported, highly efficient Philips gasifier stove. Intervention households were randomized into four different groups, three of which received different combinations of two improved stoves, while the fourth group serves as a control for the duration of the study. Diverse measurements assess different points along the causal chain linking the intervention to final outcomes of interest. The investigators assess stove use and cooking behavior, cooking emissions, household air pollution and personal exposure, health burden, and local to regional air quality. Integrated analysis and modeling will tackle a range of interdisciplinary science questions, including examining ambient exposures among the regional population, assessing how those exposures might change with different technologies and behaviors, and estimating the comparative impact of local behavior and technological changes versus regional climate variability and change on local air quality and health outcomes.

ELIGIBILITY:
Inclusion

Individual Participants:

* Classified as "rural"
* Uses biofuel as main cooking fuel source (firewood, animal waste, crop residue/sawdust)
* Uses borehole as main water source (to facilitate social network analysis linking household's knowledge and attitudes toward stoves to experience of social contacts);
* Does not have electricity (to permit possible addition of lighting intervention at a later date);
* Has a woman in household aged 18-55 and at least one child under five (since women and children are the most vulnerable to cookstove smoke and are thus the main focus of our health measures).

Clusters:

* No more than 25% classified as urban
* Accessible year-round (determined by field staff)
* Having at least 10 eligible households (in line with the participant criteria above)

Exclusion:

* Household could not be located
* Household declined to participate

Ages: 0 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 200 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Health (Biomarkers of inflammation) | At baseline
  Health indicators from blood spot samples (C-Reactive Protein, Sicam, sVCAM, serum amyloid A, Interleukin-1b, Interleukin-6, Interleukin-8, tumor necrosis factor alpha).
Health (Biomarkers of inflammation) | At 6 months
  Health indicators from blood spot samples (C-Reactive Protein, Sicam, sVCAM, serum amyloid A, Interleukin-1b, Interleukin-6, Interleukin-8, tumor necrosis factor alpha).
Health (Biomarkers of inflammation) | At 12 months
  Health indicators from blood spot samples (C-Reactive Protein, Sicam, sVCAM, serum amyloid A, Interleukin-1b, Interleukin-6, Interleukin-8, tumor necrosis factor alpha).
Health (Biomarkers of inflammation) | At 18 months
  Health indicators from blood spot samples (C-Reactive Protein, Sicam, sVCAM, serum amyloid A, Interleukin-1b, Interleukin-6, Interleukin-8, tumor necrosis factor alpha).
Height | At baseline
  Height of participants
Height | At 6 months
  Height of participants
Height | At 12 months
  Height of participants
Height | At 18 months
  Height of participants
Weight | At baseline
  Weight of participants
Weight | At 6 months
  Weight of participants
Weight | At 12 months
  Weight of participants
Weight | At 18 months
  Weight of participants
Mid-arm circumference | At baseline
  Measurement of mid-upper arm circumference of participants
Mid-arm circumference | At 6 months
  Measurement of mid-upper arm circumference of participants
Mid-arm circumference | At 12 months
  Measurement of mid-upper arm circumference of participants
Mid-arm circumference | At 18 months
  Measurement of mid-upper arm circumference of participants

SECONDARY OUTCOMES:
Personal exposure to fine particulate matter (PM2.5) | 48 hour deployment periods
  48 hour integrated personal PM2.5 concentrations from filter measurements
Personal exposure to carbon monoxide (CO) | 48 hour deployment periods
  Daily average and integrated personal CO concentrations
Kitchen area concentrations of carbon monoxide (CO) | 48 hour deployment periods
  Daily average and integrated kitchen area CO concentrations
Kitchen area concentrations of fine particulate matter (PM2.5) | 48 hour deployment periods
  48 hour integrated kitchen area PM2.5 concentrations from filter measurements
Self-reported stove usage | At baseline
  Surveys administered to respondents (primary cooks)
Self-reported stove usage | At 6 months
  Surveys administered to respondents (primary cooks)
Self-reported stove usage | At 12 months
  Surveys administered to respondents (primary cooks)
Self-reported stove usage | At 18 months
  Surveys administered to respondents (primary cooks)
Stove usage as measured by devices | Throughout data collection period, approximately 2 years.
  Continuous stove usage indicators as measured by temperature loggers on stoves

IPD SHARING:
Plan to Share IPD: No
De-identified data are available upon request.

REFERENCES:
- [Background] Dickinson KL, Kanyomse E, Piedrahita R, Coffey E, Rivera IJ, Adoctor J, Alirigia R, Muvandimwe D, Dove M, Dukic V, Hayden MH, Diaz-Sanchez D, Abisiba AV, Anaseba D, Hagar Y, Masson N, Monaghan A, Titiati A, Steinhoff DF, Hsu YY, Kaspar R, Brooks B, Hodgson A, Hannigan M, Oduro AR, Wiedinmyer C. Research on Emissions, Air quality, Climate, and Cooking Technologies in Northern Ghana (REACCTING): study rationale and protocol. BMC Public Health. 2015 Feb 12;15:126. doi: 10.1186/s12889-015-1414-1. PMID 25885780
- [Derived] Abdo M, Kanyomse E, Alirigia R, Coffey ER, Piedrahita R, Diaz-Sanchez D, Hagar Y, Naumenko DJ, Wiedinmyer C, Hannigan MP, Oduro AR, Dickinson KL. Health impacts of a randomized biomass cookstove intervention in northern Ghana. BMC Public Health. 2021 Dec 4;21(1):2211. doi: 10.1186/s12889-021-12164-y. PMID 34863138